CLINICAL TRIAL: NCT04956757
Title: Investigating the Effect of Scapula Retraction Exercises on Acromiohumeral Distance Values and Symptoms (Pain and Disability) in Patients With SPS
Brief Title: Scapula Retraction Exercises in Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Eraslan, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GO18/55
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Rotator Cuff Impingement Syndrome
Keywords: pain severity; functional status; acromiohumeral distance; shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): exercise program consists of progressive scapula retraction exercises will be applied three times a week total 24 sessions.
  Home exercise program will also advised two times a day.
  Interventions: Other: Exercise Intervention
- Control Group (No Intervention): Control group will not perform scapula retraction exercises. AHD values of the control group will be compared to intervention groups both retracted and non-retracted conditions.

INTERVENTIONS:
Other: Exercise Intervention — Scapula retraction exercises at varying shoulder abduction angles will be applied
  Arms: Intervention Group

SUMMARY:
Scapula retraction exercises are often recommended as a part of the exercise programs. The primary aim of this study is to investigate the initial effect of the scapula retraction exercises on acromiohumeral distance (AHD) at varying shoulder abduction angles and to compare asymptomatic subjects. The secondary aim of this study is to investigate the effect of scapula retraction exercises on AHD values and symptoms (pain and disability) in patients with SPS.

DETAILED DESCRIPTION:
Subacmial pain syndrome (SPS) is a common cause of shoulder pain and dysfunction in the general population. Exercise interventions is thought as a primary choice in clinical settings. Scapula retraction exercises are commonly recommended as a part of the exercise programs. Applying scapula retraction exercises at varying shoulder abduction angles could restore balance between the scapulothoracic muscles. Since the scapulothoracic muscles dynamically control subacromial space, scapula retraction exercises could further help to maintain AHD during arm elevation.

The primary aim of this study is to investigate the initial effect of the scapula retraction exercises on acromiohumeral distance (AHD) at varying shoulder abduction angles and to compare asymptomatic subjects. The secondary aim of this study is to investigate the effect of scapula retraction exercises on AHD values and symptoms (pain and disability) in patients with SPS.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* aged between 18-45
* painful arc of movement during flexion or abduction;
* positive Neer or Kennedy-Hawkins impingement signs
* pain on resisted lateral rotation, abduction or empty can test.

Exclusion Criteria:

* previous shoulder surgery;
* shoulder pain reproduced by neck movement;
* clinical signs of full-thickness RC tears; or
* adhesive capsulitis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Acromiohumeral Distance (AHD) measurement | Acromiohumeral distance values will be recorded at baseline and 8-week follow-up
  Acromiohumeral Distance will be recorded at 0°, 30°, 45°, 60° and 90° of shoulder abduction, and while they are doing scapular retraction with resistive elastic band at each shoulder position. All assessment will be recorded at baseline and at the end of the eight week rehabilitation sessions

SECONDARY OUTCOMES:
pain severity | pain severity will be recorded at baseline and 8-week follow-up
  pain severity will be assessed by using 100 millimeters Visual Analogue Scale at rest, at night and during activity.
  All patients were asked to mark their pain level that corresponds to their pain intensity on the line between "0=no pain" and "100=the worst pain imaginable".
disability status | PADI Score will be recorded at baseline and 8-week follow-up
  disability status will be assessed by using Shoulder Pain and Disability Index (SPADİ). All assessment will be recorded at baseline and at the end of the eight week treatment sessions.
  The questionnaire is scored on a 100-point scale, where 0 represents "no disabilities" and 100 represents "extreme disabilities"

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided